CLINICAL TRIAL: NCT01940822
Title: Cardiovascular Effects of Energy Drinks in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Anna Svatikova, Assistant Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 13-001918
Record Dates: First submitted 2013-09-09; First posted 2013-09-12 (Estimated); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Energy Drinks; Hemodynamics; Cardiovascular System
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Energy drink first, then placebo drink (Experimental): Participants will receive an energy drink at the first study visit, and a placebo drink at the second study visit.
  Interventions: Other: Energy Drink; Other: Placebo Drink
- Placebo drink first, then energy drink (Experimental): Participants will receive a placebo drink at the first study visit and an Energy Drink at the second study visit.
  Interventions: Other: Energy Drink; Other: Placebo Drink

INTERVENTIONS:
Other: Energy Drink
Other: Placebo Drink

SUMMARY:
This study is being done to look at the cardiovascular response, if any, to intake of commercially available energy drink. We hypothesize that energy drink consumption compared to a control drink in healthy adults alters the cardiovascular hemodynamic system.The focus of this study is to elucidate the physiological/cardiovascular response to an energy drink consumption as compared to a control drink both at rest and during stressful conditions in healthy adults.

DETAILED DESCRIPTION:
The study will collect data to determine the hemodynamic changes (magnitude of heart rate and blood pressure response) in healthy adults after consumption of an energy drink and compare these responses to those after a control drink. Study will be performed at a hospital Clinical Research Unit on two separate days; minimum 24 hours and maximum 1 month apart. Participants will be fasting 4 hours prior to the study and will be asked to abstain from caffeine and alcohol for at least 24 hours prior to initiation of this study. Baseline measurements will be obtained during and after 10 minutes of rest. After the end of baseline recordings, the subjects will be given up to 500 ml (1 can, approximately 16 fluid ounces) of caffeinated energy drink or a control drink, based on randomization. They will have 30 minutes to drink it. The second set of measurements will be obtained after an energy drink or control drink intake, using exactly the same protocol as at baseline. The second study visit, participant will receive the alternate intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and older
* Healthy subjects without known cardiovascular disease and thyroid disease
* Subjects who are on no medications (except oral contraceptive pill)
* Nonsmokers
* No prior history of caffeine sensitivity or allergy

Exclusion Criteria:

* Subjects with known cardiovascular and/or thyroid disease
* Subjects currently taking medications other than oral contraceptive pill
* Smokers
* Prior history of caffeine sensitivity or allergy
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-07; Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | Baseline, 30 minutes after consumption

SECONDARY OUTCOMES:
Change in heart rate | Baseline, 30 minutes after consumption
Change in Plasma Norepinephrine | Baseline, 30 minutes after consumption

CONTACTS AND LOCATIONS:
Overall Officials: Anna Svatikova, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Svatikova A, Covassin N, Somers KR, Somers KV, Soucek F, Kara T, Bukartyk J. A Randomized Trial of Cardiovascular Responses to Energy Drink Consumption in Healthy Adults. JAMA. 2015 Nov 17;314(19):2079-82. doi: 10.1001/jama.2015.13744. No abstract available. PMID 26547226
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials